CLINICAL TRIAL: NCT00670241
Title: A Phase 3 Study Comparing a Gel Containing Calcipotriol 50 mcg/g Plus Betamethasone 0.5 mg/g (as Dipropionate) With Tacalcitol Ointment (4 mcg/g) and Gel Vehicle, Used Once Daily in the Treatment of Psoriasis Vulgaris
Brief Title: Efficacy and Safety of Calcipotriol Plus Betamethasone Dipropionate Gel Compared With Tacalcitol Ointment and the Gel Vehicle Alone in Patients With Psoriasis Vulgaris
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LEO 80185-G21
Record Dates: First submitted 2008-04-29; First posted 2008-05-01 (Estimated); Results first posted 2011-03-08 (Estimated); Last update posted 2025-03-10 (Actual); Status verified 2015-03

CONDITIONS: Psoriasis Vulgaris
MeSH Terms: interventions — calcipotriene; Betamethasone

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator)
  Interventions: Drug: calcipotriol and betamethasone (LEO 80185 gel)
- 2 (Active Comparator)
  Interventions: Drug: Tacalcitol ointment
- 3 (Placebo Comparator)
  Interventions: Drug: LEO 80185 vehicle

INTERVENTIONS:
Drug: calcipotriol and betamethasone (LEO 80185 gel) — Once daily application
  Arms: 1
Drug: LEO 80185 vehicle — Once daily application
  Arms: 3
Drug: Tacalcitol ointment — Once daily application
  Arms: 2

SUMMARY:
This study will compare efficacy and safety of once daily treatment of calcipotriol plus betamethasone dipropionate gel (LEO 80185) with tacalcitol ointment and LEO 80185 vehicle alone in subjects with psoriasis vulgaris. Subjects will be treated for up to 8 weeks followed by an observation period of up to 8 weeks to investigate the occurence and the time to relapse and occurence of rebound after discontinuation of the investigational products. Only subjects with "controlled disease" will be considered for this observation phase of the study. "Controlled disease" is defined as "Clear" or "Almost Clear" severity category based on Investigator's global assessment (IGA).

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent to be obtained prior to any trial related procedure, including wash-out
* Clinical diagnosis of psoriasis vulgaris involving trunk and/or arms and/or legs amenable to treatment with a maximum of 100 g of LEO 80185 gel per week or 10 g per day of tacalcitol ointment
* Disease severity graded moderate, severe or very severe according to the Investigator's global assessment (IGA) of disease severity
* A minimum PASI score for extent of 2 in at least one body region (i.e.psoriasis affecting at least 10% of arms, and/or 10% of trunk, and/or 10% of legs)
* Subjects aged 18 years or above
* Either sex
* Any ethnic origin
* Attending hospital outpatient clinic or the private practice of a dermatologist

Exclusion Criteria:

* Systemic treatment with biological therapies (marketed or not marketed), with a possible effect on psoriasis vulgaris (e.g., alefacept, efalizumab, etanercept, infliximab, adalimumab) within 3 months prior to randomisation
* Systemic treatment with all other therapies than biologics, with a possible effect on psoriasis vulgaris (e.g., corticosteroids, retinoids, immunosuppressants) within 4 weeks prior to randomisation
* Systemic treatment with Vitamin D preparations above 500 IU per day
* PUVA or Grenz ray therapy within 4 weeks prior to randomization
* UVB therapy within 2 weeks prior to randomisation
* Any topical treatment of the trunk/limbs (except for emollients) within 2 weeks prior to randomisation
* Topical treatment for other relevant skin disorders on the face and flexures (e.g., facial and flexural psoriasis, eczema) with potent or very potent (WHO group III-IV) corticosteroids or vitamin D analogues within 2 weeks prior to randomisation
* Topical treatment for other relevant skin disorders on the scalp (e.g. scalp psoriasis) with very potent (WHO group IV) corticosteroids or vitamin D analogues within 2 weeks prior to randomisation
* Planned initiation of, or changes to concomitant medication that could affect psoriasis vulgaris (e.g., beta blockers, ACE inhibitors, anti-malaria drugs, lithium) during the study
* Current diagnosis of erythrodermic, exfoliative or pustular psoriasis
* Subjects with any of the following conditions present on the treatment area: viral (e.g., herpes or varicella) lesions, fungal and bacterial skin infections, parasitic infections, skin manifestations in relation to syphilis or tuberculosis, rosacea, perioral dermatitis, acne vulgaris, atrophic skin, striae atro-phicae, fragility of skin veins, ichthyosis, acne rosacea, ulcers and wounds
* Known or suspected disorders of calcium metabolism associated with hypercalcaemia
* Known or suspected severe renal insufficiency or severe hepatic disorders
* Known or suspected hypersensitivity to component(s) of the Investigational Products
* Current participation in any other interventional clinical study
* Subjects who have received treatment with any non-marketed drug substance (i.e. an agent which has not yet been made available for clinical use following registration) within the 4-week period prior to randomisation, except for biologics (3 months)
* Planned exposure to sun during the study that may affect psoriasis vulgaris
* Previously randomised to this study
* Subjects known or suspected of not being able to comply with a trial protocol (e.g. due to alcoholism, drug dependency or psychotic state)
* Females of child-bearing potential wishing to become pregnant during the study, or are breast-feeding, or not using an adequate method of contraception during the study
* Females of child-bearing potential with positive pregnancy test at Visit 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 458 (Actual)
Dates: Start 2008-04; Primary Completion 2009-02 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Langley, MD, Principal Investigator — Eastern Canada Cutaneous Research Associates Ltd.
Locations (1):
- Eastern Canada Cutaneous Research Associates Ltd., Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Clinical Trials at LEO Pharma — https://www.leopharmatrials.com/en

RESULTS

PARTICIPANT FLOW:
Groups:
- Calcipotriol Plus Betamethasone Dipropionate Gel: Calcipotriol Plus Betamethasone Dipropionate Gel for up to 8 weeks
- Tacalcitol Ointment: Tacalcitol Ointment for up to 8 weeks
- Gel Vehicle: Gel Vehicle for up to 8 weeks
Period: Overall Study
Arm/Group | Calcipotriol Plus Betamethasone Dipropionate Gel | Tacalcitol Ointment | Gel Vehicle
Started | 183 | 184 | 91
Completed | 171 | 163 | 64
Not Completed | 12 | 21 | 27

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Calcipotriol Plus Betamethasone Dipropionate Gel | Tacalcitol Ointment | Gel Vehicle | Total
Number analyzed (Participants) | 183 | 184 | 91 | 458
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 148 | 155 | 74 | 377
  >=65 years | 35 | 29 | 17 | 81
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.9 (14.3) | 51.7 (13.4) | 52.8 (14.9) | 51.6 (14.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 69 | 38 | 173
  Male | 117 | 115 | 53 | 285
Region of Enrollment [Number; unit: participants]
  Canada | 183 | 184 | 91 | 458

OUTCOME MEASURES:

1. Primary Outcome: Subjects With "Controlled Disease" ("Clear" or "Almost Clear" Disease) According to Investigator's Global Assessment of Disease Severity at Week 8
Time Frame: Week 8
Measure: Number; unit: Participants
Arm/Group | Calcipotriol Plus Betamethasone Dipropionate Gel | Tacalcitol Ointment | Gel Vehicle
Number analyzed (Participants) | 183 | 184 | 91
Participants | 73 | 33 | 5
Statistical Analysis 1: Comparison: Calcipotriol Plus Betamethasone Dipropionate Gel vs Tacalcitol Ointment; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 3.42, 95% CI 2-sided [2.05 to 5.70]

2. Secondary Outcome: Subjects With "Controlled Disease" According to the Investigator's Global Assessment of Disease Severity at Week 4
Time Frame: Week 4
Measure: Number; unit: participants
Arm/Group | Calcipotriol Plus Betamethasone Dipropionate Gel | Tacalcitol Ointment | Gel Vehicle
Number analyzed (Participants) | 183 | 184 | 91
participants | 34 | 12 | 1
Statistical Analysis 1: Comparison: Calcipotriol Plus Betamethasone Dipropionate Gel vs Tacalcitol Ointment; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 3.51, 98.33% CI 2-sided [1.46 to 8.40]

3. Secondary Outcome: The Percentage Change in PASI From Baseline to Week 8
Description: PASI is Psoriasis Area and Severity Index and is based on the investigator's assessment of extent and severity of the disease. It can range from 0 (best) to 64.8 (worst).
Time Frame: Baseline, Week 4 and 8
Measure: Number; unit: Percent change in PASI score
Arm/Group | Calcipotriol Plus Betamethasone Dipropionate Gel | Tacalcitol Ointment | Gel Vehicle
Number analyzed (Participants) | 183 | 184 | 91
Percent change in PASI score | -57.0 | -41.9 | -17.9
Statistical Analysis 1: Comparison: Calcipotriol Plus Betamethasone Dipropionate Gel vs Tacalcitol Ointment; Test type: Superiority or Other; p < 0.001, ANOVA; Mean Difference (Final Values) = -14.7, 98.33% CI 2-sided [-22.6 to -6.90]

4. Secondary Outcome: Subjects With Relapse During the Study
Description: Among subjects with controlled disease at week 8 relapse was defined as PASI exceeding the baseline PASI value minus 50% of the reduction in PASI obtained from the baseline visit to the last on-treatment visit
Time Frame: Week 8-16
Measure: Number; unit: participants
Arm/Group | Calcipotriol Plus Betamethasone Dipropionate Gel | Tacalcitol Ointment | Gel Vehicle
Number analyzed (Participants) | 67 | 31 | 5
participants | 28 | 7 | 3

5. Secondary Outcome: Subjects With Rebound During the Study
Time Frame: Week 8-16
Measure: Number; unit: participants
Arm/Group | Calcipotriol Plus Betamethasone Dipropionate Gel | Tacalcitol Ointment | Gel Vehicle
Number analyzed (Participants) | 67 | 31 | 5
participants | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Calcipotriol Plus Betamethasone Dipropionate Gel | Tacalcitol Ointment | Gel Vehicle
Serious Adverse Events (participants affected / at risk) | 0/182 | 4/184 | 1/91
Other Adverse Events (participants affected / at risk) | 25/182 | 28/184 | 10/91
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Calcipotriol Plus Betamethasone Dipropionate Gel (N=182) | Tacalcitol Ointment (N=184) | Gel Vehicle (N=91)
Arrhythmia (Cardiac disorders) | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Calcipotriol Plus Betamethasone Dipropionate Gel (N=182) | Tacalcitol Ointment (N=184) | Gel Vehicle (N=91)
Nasopharyngitis (Infections and infestations) | 11 | 6 | 1
Upper respiratory tract infection (Infections and infestations) | 8 | 10 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 6 | 13 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No